CLINICAL TRIAL: NCT04234711
Title: Sutureless Technique and Conventional Repairs for Total Anomalous Pulmonary Venous Connection: an Observational Study by Chinese Heart Centers
Brief Title: Sutureless Technique and Conventional Repairs for Total Anomalous Pulmonary Venous Connection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20190505
Record Dates: First submitted 2020-01-12; First posted 2020-01-21 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Total Anomalous Pulmonary Venous Connection
Keywords: TAPVC; Surgical strategy; PVO; outcomes
MeSH Terms: conditions — Scimitar Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Common pulmonary vein tissue for histopathology of abnormal vein
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional surgical group: Patients with total pulmonary venous connection undergo conventional surgical repair
  Interventions: Procedure: Surgical strategy
- Sutureless surgical group: Patients with total pulmonary venous connection undergo sutureless surgical repair
  Interventions: Procedure: Surgical strategy

INTERVENTIONS:
Procedure: Surgical strategy — To compare the efficacy between conventional repair and sutureless technique for total anomalous pulmonary venous connection

SUMMARY:
The purpose of this study is to evaluate the efficacy of conventional repair and sutureless surgical repair of total anomalous pulmonary venous connection.

DETAILED DESCRIPTION:
An observational, non-randomized multi-center study is proposed to compare the efficacy between conventional repair and sutureless technique for total anomalous pulmonary venous connection. Subjects will be enrolled at Guangdong Provincial People's Hospital (GPPH) and three to five participating hospitals. All clinical interventions will follow the participating hospital's standard of care. Informed consent will be obtained from all study participants before study enrollment. After undergoing their surgical repairs, study participants will be followed up at 1, 3, 6 and 12 months after initial surgery and annually thereafter. All preoperative and postoperative medical records data will be submitted to a centralized database at GPPH through a secure online research platform.

Baseline and post-operative (6 months) assessments will include a history and physical examination, a quality of life survey, physical examinations, liver and kidney function assessments, serum brain natriuretic peptide (BNP), echocardiography and electrocardiography. Besides, a small amount of common pulmonary vein tissue may be required for hematein and eosin staining.

ELIGIBILITY:
Inclusion Criteria:

1. Infants and neonates who are diagnosed with TAPVC
2. Infants and neonates who undergo initial surgical repair for TAPVC.

Exclusion Criteria:

1. Concommitant diagnoses including functional single ventricular, double outlet right ventricle, tricuspid atresia, pulmonary atresia, or transposition of the great arteries.
2. Older than 1-year-old.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates and infants undergoing initial operation for total anomalous pulmonary venous connection in the participating hospitals of this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-02-20 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of postoperative pulmonary venous obstruction (PVO) | 2 years
  in anastomosis or arborizations of pulmonary veins
Mortality rate | 2 years
  all causes and surgical repair related

SECONDARY OUTCOMES:
The scores of postoperative quality of life: rating scale | 2 years
  Fill the rating scale through telephone or other communication
Change in resting oxygen saturation | 2 years
  Answer question through telephone or other communication
Value of tricuspid annular plane systolic excursion | 2 years
  Measured by echocardiology from follow-up
Development of all kinds of arrhythmia | 2 years
  Measured by electrocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhuang, M.D., Ph D., Study Director — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No